CLINICAL TRIAL: NCT01043068
Title: A Pilot Study: The Effect of Cancer Pain Management Protocol on Hospitalized Cancer Patients
Brief Title: The Effect of Cancer Pain Management Protocol on Hospitalized Cancer Patients: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Principal Investigator, Sang Myung Woo, MD, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAPAM-1
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Cancers, Pain
Keywords: cancer pain; opioid; guideline
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pain control (Experimental): Interventions based on published pain guideline. The interventions consisted of the following: (1) nursing pain assessment of current pain, worst pain, pain relief, and acceptability of pain; (2) feedback to guide analgesic prescribing by physician.
  Interventions: Drug: Cancer pain management

INTERVENTIONS:
Drug: Cancer pain management — Interventions based on published pain guideline. The interventions consisted of the following: (1) nursing pain assessment of current pain, worst pain, pain relief, and acceptability of pain; (2) feedback to guide analgesic prescribing by physician.

SUMMARY:
The purpose of this study was to prospectively evaluate the effect of cancer pain management protocol on hospitalized cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient with the somatic and/or visceral pain having an untreated intensity greater than 3 on a 10 cm visual analog scale (VAS; 0 = no pain, 10 = unbearable pain)over the week prior to enrollment
* A minimum age of 18 years

Exclusion Criteria:

* Opioid intolerance
* No longer treatment for their underlying disease.
* Intracerebral primary or metastatic lesion
* Impaired sensory or cognitive function
* Pregnant or lactating woman
* Women of child bearing potential not using a contraceptive method
* Sexually active fertile men not using effective birth control during medication of study drug and up to 6 months after completion of study drug if their partners are women of child-bearing potential
* Any patients judged by the investigator to be unfit to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction in pain scores | Jan 2010 - October 2010

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Kim, Prof, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea